CLINICAL TRIAL: NCT03180307
Title: A Phase 3, Randomized, Single Dose, Open-Label Study to Investigate the Safety and Efficacy of OTL38 Injection (OTL38) for Intra-operative Imaging of Folate Receptor Positive Ovarian Cancer
Brief Title: OTL38 for Intra-operative Imaging of Folate Receptor Positive Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: On Target Laboratories, LLC (Industry)
Collaborators: SynteractHCR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OTL-2016-OTL38-006
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Pafolacianine; Injections; Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- no fluorescent imaging (Sham Comparator): Patient injected with OTL38, but does not undergo fluorescent imaging
  Interventions: Drug: OTL38; Procedure: laparotomy
- near infrared imaging arm (Experimental): Patient injected with OTL38 and undergoes near infrared imaging
  Interventions: Drug: OTL38; Device: near infrared camera imaging system; Procedure: laparotomy

INTERVENTIONS:
Drug: OTL38 — 0.025 mg/kg of OTL38 in 250ml dextrose 5% in water (D5W) infused intravenously over 60 minutes
  Other Names: OTL38 for Injection
Device: near infrared camera imaging system — Infrared imaging used to excite OTL38 for fluorescence
  Other Names: Near IR imaging
  Arms: near infrared imaging arm
Procedure: laparotomy — primary surgical cytoreduction, interval debulking, or recurrent ovarian cancer surgery

SUMMARY:
This is a phase 3, randomized, multi-center, single dose, open label, pivotal study in patients diagnosed with, or with high clinical suspicion of, ovarian cancer scheduled to undergo primary surgical cytoreduction, interval debulking, or recurrent ovarian cancer surgery.

DETAILED DESCRIPTION:
The Phase 3 study is to confirm the efficacy of OTL38 in combination with fluorescent light to detect additional Folate Receptor-positive (FR+) ovarian cancer lesions not detected by palpation and visualization under normal light in patients with FR+ ovarian cancer scheduled to undergo primary surgical cytoreduction, interval debulking, or recurrent ovarian cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age and older
* Have a primary diagnosis, or at high clinical suspicion, of primary ovarian cancer (of epithelial type), planned for primary surgical cytoreduction, interval debulking, or have recurrent ovarian cancer surgery, and:

  * Who are scheduled to undergo laparotomy for the debulking surgery OR
  * Who are scheduled to undergo laparoscopy and pre-authorized to undergo laparotomy for the debulking surgery if cancer is detected on the laparoscopy
* A negative serum pregnancy test at Screening followed by a negative urine pregnancy test on the day of surgery or day of admission for female patients of childbearing potential
* Female patients of childbearing potential or less than 2 years postmenopausal agree to use an acceptable form of contraception from the time of signing informed consent until 30 days after study completion
* Ability to understand the requirements of the study, provide written informed consent for participation in the study and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments

Exclusion Criteria:

* Previous exposure to OTL38
* Known FR-negative ovarian cancer
* Planned surgical debulking via laparoscopy or robotic surgery, with no intent of laparotomy.
* Patients with known ovarian cancer miliary disease determined preoperatively to be inoperable.
* Any medical condition that, in the opinion of the investigators, could potentially jeopardize the safety of the patient
* History of anaphylactic reactions
* History of allergy to any of the components of OTL38, including folic acid
* Pregnancy or positive pregnancy test
* Clinically significant abnormalities on electrocardiogram (ECG)
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Impaired renal function defined as eGFR< 50 mL/min/1.73m2
* Impaired liver function defined as values > 3x the upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin.
* Known Stage IV ovarian cancer with brain metastases
* Received an investigational agent in another clinical trial within 30 days prior to surgery
* Known sensitivity to fluorescent light

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janos Tanyi, MD, Principal Investigator — University of Pennsylvania
Locations (11):
- United States (10):
  - The Mayo Clinic - Phoenix, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - City of Hope Medical Center, Duarte, California
  - University of CA at Irvine Chao Cancer Center, Orange, California
  - Moffitt Cancer Center, Tampa, Florida
  - Karmanos Cancer Institutes, Detroit, Michigan
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Kettering Medical Center, Kettering, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanyi JL, Randall LM, Chambers SK, Butler KA, Winer IS, Langstraat CL, Han ES, Vahrmeijer AL, Chon HS, Morgan MA, Powell MA, Tseng JH, Lopez AS, Wenham RM. A Phase III Study of Pafolacianine Injection (OTL38) for Intraoperative Imaging of Folate Receptor-Positive Ovarian Cancer (Study 006). J Clin Oncol. 2023 Jan 10;41(2):276-284. doi: 10.1200/JCO.22.00291. Epub 2022 Sep 7. PMID 36070540

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: OTL38 Injection and Near Infrared Imaging: Patient injected with OTL38 and undergoes near infrared imaging.
  Drug: OTL38 0.025 mg/kg of OTL38 in 250ml dextrose 5% in water (D5W) infused intravenously over 60 minutes
  Other Names:
  OTL38 for Injection Device: near infrared camera imaging system Infrared imaging used to excite OTL38 for fluorescence
  Other Names:
  Near IR imaging Procedure/Surgery: laparotomy primary surgical cytoreduction, interval debulking, or recurrent ovarian cancer surgery
- Sham Comparator: OTL38 Injection and No Fluorescent Imaging: Patient injected with OTL38, but does not undergo fluorescent imaging.
  Drug: OTL38 0.025 mg/kg of OTL38 in 250ml dextrose 5% in water (D5W) infused intravenously over 60 minutes
  Other Names:
  OTL38 for Injection Procedure/Surgery: laparotomy primary surgical cytoreduction, interval debulking, or recurrent ovarian cancer surgery
Period: Overall Study
Arm/Group | Experimental: OTL38 Injection and Near Infrared Imaging | Sham Comparator: OTL38 Injection and No Fluorescent Imaging
Started | 134 | 6
Safety Analysis Set (All subjects received study drug prior to randomization. A total of 150 subjects received study drug, 10 of which were not randomized to either arm. These 10 subjects withdrew to the study prior to randomization but are included in the Safety Analysis Set.) | 134 | 16
Full Analysis Set/ Intent to Image Set | 134 | 0
Per Protocol Analysis Set | 106 | 0
Pharmacokinetic Analysis Set | 122 | 6
Completed | 128 | 6
Not Completed | 6 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 1 | 0
Not completed — Majority of which were disease too extensive and camera not used | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: OTL38 Injection and Near Infrared Imaging | Sham Comparator: OTL38 Injection and No Fluorescent Imaging | Total
Number analyzed (Participants) | 134 | 6 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.91) | 62.8 (21.77) | 60.8 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 6 | 140
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 2 | 17
  Not Hispanic or Latino | 116 | 4 | 120
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 114 | 5 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Patient Level
Description: Percentage of patients with at least one evaluable FR+ ovarian cancer lesion confirmed by central pathology (Standard of truth) that was detected using the combination of OTL38 and fluorescent light but not under normal light or palpation (Full Analysis Set)
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Full Analysis Set: Patients exposed to OTL38 and who were randomly assigned to undergo NIR fluorescent imaging (OTL38+imaging) and who:
  * Were evaluated under both normal light and NIR fluorescent light imaging
  * Had central pathology and histology confirmation for at least one FR+ ovarian cancer lesion detected under normal light or NIR fluorescent light imaging
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 134
percentage of participants | 26.9 [19.6 to 35.2]

2. Secondary Outcome: Patient False Positive Rate
Description: False Positive Rate at the patient level (FPRp) will be a major secondary efficacy endpoint and is defined as the percentage of women who underwent both normal light and fluorescent light (Intent-to-Image Set)
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 134
percentage of participants | 20.2 [13.7 to 28.0]

ADVERSE EVENTS:
Time Frame: Incidence rates of treatment-emergent AEs (TEAEs), SAEs, and Adverse Device Effects (ADEs) Visit 1 (screening) through Visit 4 (28 days +/- 7 days).
Description: The "Other Adverse Events" table captures all drug-related treatment-emergent adverse events reported at or above the frequency threshold for reporting.
Groups:
- Safety Analysis Set: The Safety Analysis Set includes all subjects who received any amount of study drug.
Arm/Group | Safety Analysis Set
All-Cause Mortality (participants affected / at risk) | 2/150
Serious Adverse Events (participants affected / at risk) | 22/150
Other Adverse Events (participants affected / at risk) | 34/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Analysis Set (N=150)
Septic shock (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Postoperative wound infection (Immune system disorders) | 1
Sepsis (Infections and infestations) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 3
Anastomotic leak (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Vaginal cuff dehiscence (Injury, poisoning and procedural complications) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Analysis Set (N=150)
Nausea (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03180307/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT03180307/SAP_001.pdf